CLINICAL TRIAL: NCT03812406
Title: Comparison Between French Ambulatory Cesarean Section to The Misgav-Ladach Technique - Double Blind Randomized Controlled Trial
Brief Title: Comparison of FAUCS vs. Misgav Ladach
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bnai Zion Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FAUCS
Record Dates: First submitted 2018-12-19; First posted 2019-01-23 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2018-12

CONDITIONS: Pain, Postoperative; Ambulation Difficulty
Keywords: cesarean
MeSH Terms: conditions — Pain, Postoperative; Mobility Limitation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FAUCS (Experimental): Patients undergoing a cesarean section using the FAUCS technique
  Interventions: Procedure: French Abulatory Cesrean Section
- Control (Active Comparator): Patients undergoing a cesarean section using the traditional (Misgav-Ladach) technique
  Interventions: Procedure: Misgav-Ladach

INTERVENTIONS:
Procedure: French Abulatory Cesrean Section — A cesarean section performed according to the FAUCS technique
  Arms: FAUCS
Procedure: Misgav-Ladach — A cesarean section performed according to the Misgav Ladach technique
  Arms: Control

SUMMARY:
This study aims to compare two techniques for performing a cesarean delivery: Misgav Ladach versus French Ambulatory Cesarean Section (FAUCS). The second techniques has been claimed to reduce post-operative pain, the need for analgesics, and reduce the time for ambulation. Such comparison has not been done so far, and this study will examined if indeed the FAUCS techniques offers any advantages.

DETAILED DESCRIPTION:
The FAUCS technique for performing a cesarean section has been described by a French group several years ago, and is claimed to reduce postoperative pain and increase ambulation. With this technique, after making the transverse skin incision, the fascia is opened vertically and to the left of the linea alba. The left rectus abdominis muscle is then pushed laterally, and the abdominal cavity is entered. The uterine incision in performed as usual. Due to the reduced incision size, a special spatula is used to facilitate extraction of the fetal head in some cases. No urinary catheter is used during or after the operation, and fluid administration is restricted during the procedure. The patient is encouraged to get out of bed 3-4 hours post surgery. This technique for performing a cesarean section will be compared with the traditional (Misgav Ladach technique) in terms of post-operative pain, need for analgesics, ambulation, neonatal outcome, and perioperative complications.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for a cesarean section
* term pregnancy: 37-42 weeks
* singleton pregnancy
* age 18 and above
* patients capable of signing an informed consent

Exclusion Criteria:

* multiple pregnancy
* emergency cesarean
* previous 3 cesareans and above
* placenta accreta
* uterine myomas in the lower segment
* fetal growth restriction
* fetal anemia
* preeclampsia
* women scheduled for general anesthesia

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 120 (Estimated)
Dates: Start 2018-08-19 (Actual); Primary Completion 2019-08-19 (Estimated); Study Completion 2019-09-19 (Estimated)

PRIMARY OUTCOMES:
Composite maternal adverse outcome | 24 hours post surgery
  The rate of women with a composite maternal adverse outcome, defined as at least one of the following: Visual Analogue Scale score >6 (scale of 1-10, 1 being a very mild pain, 10 being the worst pain imagineable) at 3-4 hours post surgery, inability to ambulate 3-4 hours post surgery, and QoR15 (Quality of Recovery) score < 90 (range 0 to 150, 150 being the best recovery after surgery) at 24 hours post surgery

SECONDARY OUTCOMES:
Length of surgery | 24 hours
  The duration of surgery (in minutes) from incision until closure.
Blood loss (ml) during surgery | 24 hours
  The estimated volume of blood (in ml) lost during surgery
Birthweight | immediately after birth
  The weight (grams) of the neonate immediately after birth
Cord pH | immediately after birth
  The pH measured in a blood sample from the umbilical artery
Birth trauma | 24 hours
  The rate of birthtrauma in diagnosed in the neonate (shoulder dystocia, fracture, cerebral hemorrhage, cephalhematoma, etc.)

CONTACTS AND LOCATIONS:
Locations (1):
- Bnai-Zion Medical Center, Haifa, Israel

REFERENCES:
- [Derived] Sagi S, Bleicher I, Bakhous R, Pelts A, Talhamy S, Caspin O, Sammour R, Sagi-Dain L. Comparison between the modified French AmbUlatory Cesarean Section and standard cesarean technique-a randomized double-blind controlled trial. Am J Obstet Gynecol MFM. 2023 Jul;5(7):100910. doi: 10.1016/j.ajogmf.2023.100910. Epub 2023 Feb 23. PMID 36828283